CLINICAL TRIAL: NCT03894072
Title: Effect of High Flow Humidified Oxygen on Non-ventilated Lung During Thoracic Surgery: a Cross-over Study Compared With Conventional CPAP (Continuous Positive Airway Pressure)
Brief Title: HFHO vs CPAP During Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Prasert Sawasdiwipachai, Associate professor, Mahidol University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Si066/2019
Record Dates: First submitted 2019-03-27; First posted 2019-03-28 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Hypoxaemia During Surgery; Lung Hyperinflation
Keywords: High flow oxygen device, HFHO, CPAP, One-lung ventilation
MeSH Terms: conditions — Microcephaly, Primary Autosomal Recessive, 6

STUDY DESIGN:
Intervention Model Description: HFHO-CPAP CPAP-HFHO
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFHO-CPAP (Active Comparator): This group will have HFHO before CPAP
  Interventions: Device: CPAP; Device: HFHO
- CPAP-HFHO (Active Comparator): This group will have CPAP and then HFHO
  Interventions: Device: CPAP; Device: HFHO

INTERVENTIONS:
Device: CPAP — Conventional CPAP
  Other Names: Mallinkrodt CPAP
Device: HFHO — A device that can provide heated humidified oxygen up to 30-60 liter per minute, FiO2 (fraction of inspired oxygen) 0.21-0.95
  Other Names: Optiflow, Airvo

SUMMARY:
A single institutional cross-over study design to compare between high flow humidified oxygen (HFHO) device versus conventional CPAP for non-ventilated lung during thoracic surgery.

DETAILED DESCRIPTION:
The investigators hypothesize that HFHO may be an alternative tool to supply oxygen to non-ventilated lung during one lung ventilation. CPAP can improve oxygenation at a cost of lung hyperinflation which is an unwanted condition during thoracic surgery especially the video-assisted one.

Recruiting adult patients who undergo lung surgeries that requires one-lung ventilation. Exclusion criteria include the followings:-

1. Emergency case.
2. Patients with severe COPD(Chronic Obstructive Pulmonary Diseases).
3. Patients with moderate baseline hypoxemia (SpO2 < 90% on room air).
4. Patients with severe hemoptysis.
5. Patients with upper or lower airway abnormalities.
6. Patients undergo pulmonary lavage.
7. Patients with known pulmonary hypertension.
8. Patients with known pulmonary/tracheobronchial infections.
9. Patients with suspected difficult airway.
10. Patients with BMI over 35.
11. Pregnant patients.

Following a standard anesthetic practice. All participants will receive an intravenous based anesthetic with or without regional blocks. The appropriate sized double lumen endobronchial tube will be placed and fiberoptic bronchoscope is used to verify a proper position. Patient will also get an arterial line for frequent ABG (Arterial Blood Gases) samplings.

Computer generated randomization will divide patients into 2 groups. Baseline ABG will be drawn. After one lung ventilation commenced for 20 minutes, the 2nd ABG will be drawn, the surgeon who was blinded to the intervention will evaluate the quality of lung collapse using 5-point Likert scale. Then, patients will either receive a CPAP or HFHO (depends on randomization) for 20 minutes. Up on 1st intervention completion, the 3rd ABG and lung collapse evaluation will be performed.

Following the first intervention, the non-ventilated lung will be suctioned out and wait for 20 minutes. Another ABG will be sampled at this point.

The patient will receive the 2nd alternative intervention (CPAP or HFHO- depend on their randomization) for 20 minutes. The final ABG and lung collapse evaluation will be performed.

If any severe hypoxemia/ hypercarbia and marked violation of protocol occurs. Patients will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* All adult > 18 years of age undergoes lung surgeries that required one-lung ventilation

Exclusion Criteria:

* emergency case
* severe COPD
* moderate baseline hypoxemia
* pulmonary hypertension
* difficult upper/lower airway
* BMI > 35
* severe pneumonia
* bronchial lavage
* massive hemoptysis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with improved oxygenation. | 20 minutes
  Improvement of gas exchanges by arterial blood gases

SECONDARY OUTCOMES:
Quality of lung collapsed. | 20 minutes
  Lung collapse quality by surgeon using 5-point Likert scale where 5 = very good, 4= good, 3 = acceptable, 2 = poor and 1= very poor

CONTACTS AND LOCATIONS:
Overall Officials: Prasert Sawasdiwipachai, MD, Principal Investigator — Mahidol University
Locations (1):
- Department of Anesthesiology, Faculty of Medicine, Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided